CLINICAL TRIAL: NCT04679480
Title: A Prospective, Open, Single-arm, Single Center, Phase II Trial to Assess the Efficacy of Anti-PD1 Antibody in Combination With Pulsed Hedgehog Inhibitor in Advanced Basal Cell Carcinoma.
Brief Title: Anti-PD1-antibody and Pulsed HHI for Advanced BCC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Reinhard Dummer (Other)
Collaborators: Sanofi (Industry); Sun Pharmaceutical Industries Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Reinhard Dummer, Prof. Dr. med, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGZ-2018-12355
Record Dates: First submitted 2020-12-03; First posted 2020-12-22 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — cemiplimab; sonidegib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Investigational product: a combination of an anti-PD1 antibody (Cemiplimab) and a HHI (Sonidegib).
  Cemiplimab will be supplied as a liquid in a sterile, single-use 10 ml vial. Each vial will contain a volume of 7ml at a concentration of 50mg/ml. Cemiplimab will be prepared for infusion at the trial site and administered as a flat 350mg dose in 100ml sodium chloride 0.9% as an IV infusion over approximately 30 minutes (±10 minutes) in an outpatient setting. Each patient's dose will be administered as a flat 350mg dose in every 3 weeks, starting from week 2 of the trial.
  The Hedgehog Inhibitor used for the trial will be Sonidegib. Sonidegib is a white 200mg capsule, orally administered once daily. Sonidegib will be administered in a 2 week cycle every 4 weeks (pulsed therapy: 2 weeks on, 2 weeks off), starting from week 0 of the trial.
  Interventions: Drug: Cemiplimab Injection [Libtayo]

INTERVENTIONS:
Drug: Cemiplimab Injection [Libtayo] — Investigational product: a combination of an anti-PD1 antibody (Cemiplimab) and a HHI (Sonidegib).
  Cemiplimab will be supplied as a liquid in a sterile, single-use 10 ml vial. Each vial will contain a volume of 7ml at a concentration of 50mg/ml. Cemiplimab will be prepared for infusion (as described in SmPC (Fachinformation Swissmedic) Libtayo, see Appendix) at the trial site and administered as a flat 350mg dose in 100ml NaCl 0.9% as an IV infusion over approximately 30 minutes (±10 minutes) in an outpatient setting. Each patient's dose will be administered as a flat 350mg dose in every 3 weeks, starting from week 2 of the trial.
  The Hedgehog Inhibitor used for the trial will be Sonidegib. Sonidegib is a white 200mg capsule, orally administered once daily. Sonidegib will be administered in a 2 week cycle every 4 weeks (pulsed therapy: 2 weeks on, 2 weeks off), starting from week 0 of the trial.
  Other Names: Sonidegib

SUMMARY:
The purpose of this study is to evaluate the tumour response, safety and induction of immune response in patients with advanced BCC treated with a combination of anti-PD1 antibody and pulsed hedgehog inhibitor.

DETAILED DESCRIPTION:
A prospective, open, single-arm, single center, phase II trial to assess the efficacy of anti-PD1 antibody in combination with pulsed Hedgehog inhibitor in advanced Basal Cell Carcinoma.

20 patients with advanced BCC will be included in the trial. No blinding or randomization will be conducted in this open label, non-randomized clinical trial. All of the patients will receive the investigative treatment (combination of anti-PD1 antibody and pulsed HHI therapy). The tumor response will be evaluated comparing tumour size at baseline, at each assessment, and 26 weeks after treatment initiation.

The study duration from screening visit to the End of Study visit is 32 weeks with a Follow-Up 1 Visit at week 28 and Follow-Up 2 Visit at week 32. The duration of the translational part (secondary objectives) of the study is up to 24 months.

If the best response any time at week 26 is partial response, patients will be offered to continue at least one of the study drugs until complete response or until a maximum of 2 years. The evaluation during this period will correspond to the standard of care with laboratory tests at each follow up and imaging every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Histologically or cytologically confirmed advanced BCC, defined as: a) metastasized BCC, b) locally advanced BCC, not suitable for surgical or radio-therapeutic treatment c) multiple BCCs (>5) d) BCC >10mm; not suitable for surgery or radiotherapy
* Subjects must have an evaluable disease as measured by Immune-related Response criteria, or PERSIST (PET response criteria in solid tumours) criteria in patients with metastatic BCCs without cutaneous lesions.
* Subjects (males and females) aged ≥ 18 years
* Adequate organ function (hematologic, renal, hepatic), as assessed by the study physician. Deviations of the following parameters are allowed upon decision of the investigator in case that these are not considered to be of clinical relevance and/or don't represent organ dysfunction or correspond to allowed comorbidities as specified in section 7.1:
* Absolute neutrophil count >1.5 x 109/l
* Hemoglobin >9 g/dL
* Platelets ≥ 100 x 109/l
* Serum total bilirubin <1.5 x Upper limit of normal (ULN) (or ≤3x ULN, if liver metastases).
* Alanine transaminase (ALT) and Aspartate transaminase (AST) < 3 x ULN or <5 ULN if liver metastases are present
* Patients with Gilbert's Disease and total bilirubin up to 3x ULN may be eligible after communication with and approval from the medical monitor
* Alkaline phosphatase (ALP) ≤2.5x ULN (or ≤5x ULN, if liver or bone metastases)
* Serum creatinine < 2 x ULN
* Creatine phosphokinase (CPK) (also known as creatine kinase (CK)) elevation ≤ grade 2
* Eastern Cooperative Oncology Group (ECOG) ≤2
* Negative pregnancy test in women of childbearing potential
* Anticipated life expectancy >12 weeks

Exclusion Criteria:

* History of documented allergic reactions or acute hypersensitivity reaction attributed to antibody treatments
* Patients with allergy or hypersensitivity to Cemiplimab or to any of the excipients of Libtayo. Specifically, because of the presence of trace components in Cemiplimab, patients with allergy or hypersensitivity to doxycycline or tetracycline are excluded.
* Patients with allergy or hypersensitivity to Sonidegib or to any of the excipients of Odomzo.
* Patients with a history of solid organ transplant (patients with prior corneal transplants may be allowed to enrol after discussion with and approval from the medical monitor)
* Receipt of live vaccines (including attenuated) within 30 days of first study treatment or patient unwilling not to receive them during the treatment and for up to 5 half-lives after the last dose of Cemiplimab
* Known of suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, due to language problems, psychological disorders, social conditions or dementia
* Currently receiving treatment with another investigational device or study drug, or <28 days since ending treatment with another investigational device or study drug
* Any anticancer treatment other than radiation therapy (chemotherapy, targeted systemic therapy, imiquimod, photodynamic therapy), investigational or standard of care, within 30 days of the initial administration of Cemiplimab or planned to occur during the study period
* Prior treatment with an agent that blocks the PD-1/PD-L1 pathway
* Prior treatment with other systemic immune-modulating agents within fewer than 28 days prior to the first dose of Cemiplimab. Prior treatment with imiquimod or other topical or intralesional immune modulators will not be exclusionary
* Female subject is pregnant or breast-feeding, or planning to become pregnant or breast-feed, or unwilling to use acceptable method(s) of effective contraception during study treatment and during 20 months after the last dose of Sonidegib; and during 6 months (4 in case of breast-feeding) after the last dose of Cemiplimab in case of a Cemiplimab monotherapy (in case of continuation of treatment as detailed in section 6.1)
* Male subject is planning to procreate, donate Semen, or unwilling to use acceptable method(s) of effective contraception during study treatment and during 6 months after the last dose of Sonidegib or Cemiplimab
* Subject is unwilling to renounce to blood spending during the treatment and during 20 months after the last dose of Sonidegib.
* Subject is unwilling to renounce to any elective surgery during the treatment period and for at least 30 days after the administration of the study drug
* Autoimmune diseases, requiring immunosuppressive systemic corticosteroid doses (10mg prednisone or equivalent), during trial participation or within 4 weeks prior to the first treatment dose. Patients who require brief courses of systemic corticosteroids (eg, as prophylaxis for imaging studies due to hypersensitivity to contrast agents) are not excluded. The following are not exclusionary: vitiligo, childhood asthma that has resolved, type 1 diabetes, residual hypothyroidism that required only hormone replacement, or psoriasis that does not require systemic treatment.
* Impaired cardiac function or clinically significant heart disease, including any of the following:
* Angina pectoris within 3 months
* Acute myocardial infarction within 3 months
* Other clinically significant heart disease (as evaluated by study physician)
* Patients, who are receiving treatment with medications that are known to be strong inhibitors or inducers of CYP3A4/5 or drugs, metabolized by CYP2B6 or CYP2C9 that cannot be discontinued prior to study entry and for duration of the study. Medications, that are strong CYP3A4/5 inhibitors should be discontinued for at least 2 days, and strong CYP3A4/5 inducers for at least 1-week prior initiating HHI
* Other anti-cancer treatment (except for topical therapies, such as cryotherapy, for skin lesions other than aBCC) within 30 days to treatment start
* Uncontrolled infection or active infection requiring therapy, including human immunodeficiency virus (HIV)-1 or HIV-2, hepatitis B virus (HBV), or hepatitis C virus (HCV)
* Previous enrolment into the current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Concurrent malignancy other than aBCC and/or history of malignancy other than aBCC within 3 years of date of first planned treatment dose, except for:
* Tumours with negligible risk of metastasis or death (such as cutaneous squamous cell carcinoma, low-risk early stage prostate adenocarcinoma or other tumours, upon decision of study physician)
* Patients with hematologic malignancies, upon decision of study physician
* Untreated brain metastasis(es) that may be considered active. Patients with previously treated brain metastases may participate provided that the lesion(s) is (are) stable (without evidence of progression for at least 6 weeks on imaging obtained in the screening period), and there is no evidence of new or enlarging brain metastases, and the patients do not require any immunosuppressive doses of systemic corticosteroids for management of brain metastasis(es) within 28 days of the first dose of Cemiplimab.
* History of pneumonitis within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Best response any time between the treatment start and 26 weeks after the initiation of the treatment. | At baseline, each assessment and the week 26.
  The response will be assessed according to the Immune-response Criteria (Appendix) in all patients with cutaneous lesions as: complete response, partial response, stable disease or progressive disease. The best response documented between treatment start and week 26 will be considered "best response". In case of metastatic BCC without cutaneous lesions at screening, the primary outcome will be assessed using PET/CT imaging according to the PERCIST criteria every 12 weeks from treatment start.
  In patient withdrawn from the trial before week 26, the last tumour assessment will be used for evaluation of primary outcome. For patients withdrawn from the study a full body physical examination and laboratory results will be performed prior to withdrawal, unless refused by the patient.

SECONDARY OUTCOMES:
Tumour response at 26 weeks after the initiation of the treatment | 26 weeks after the initiation of the treatment
  The secondary outcome tumour response at 26 weeks after treatment initiation will be evaluated at week after treatment start, or at the end of treatment, whichever comes first.
Detection of histologic changes in the tumour in patients with biopsy-assessable tumours | Histologic changes will be compared in the biopsies taken at baseline, week 2, week 26, and, if applicable, week 4 and week 12.
  The following histologic changes in the tumor will be measured:
  * CD4 Infiltration
  * CD8 Infiltration
  * TREG FOXP3 infiltration
Evaluation of the changes in immunogenicity of the tumour and tumour microenvironment in patients with biopsy-assessable tumours | Immunogenicity will be compared in the biopsies taken at baseline, week 2, week 26, and, if applicable, week 4 and week 12.
  The following changes in immunogenicity will be evaluated:
  * MHC-I expression
  * TAP-I expression
  * TAP-II expression
  * B-Catenin expression
  * PD-1 expression
  * PD-L1 expression
  * CD-200 expression
  * SOX-9 expression
  * BCL-2 expression

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Dummer, Prof., Principal Investigator — University Hospital Zurich, Clinic of Dermatology
Locations (1):
- University Hospital Zurich, Clinic of Dermatology, Zurich, Switzerland